CLINICAL TRIAL: NCT03483337
Title: Quantitative Imaging Tools to Derive DW-MRI Oncological Biomarkers
Brief Title: New MRI Biomarkers in Head and Neck Cancers
Status: Recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 18-063
Record Dates: First submitted 2018-03-19; First posted 2018-03-30 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Head and Neck Cancer; Thyroid Cancer
Keywords: (DW)-MRI; oncological biomarkers; metastatic; recurrent; 18-063
MeSH Terms: conditions — Head and Neck Neoplasms; Thyroid Neoplasms; Neoplasm Metastasis; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- recurrent or metastatic head and neck cancer patients: Patients will be imaged on a 1.5 T or 3 T MR scanner. Patients will receive a test-retest DWI scan in on session prior to start of treatment. Patients who will be receiving radiation therapy treatment at Memorial Sloan Kettering's main campus, will also be imaged weekly during their course of treatment.
  Interventions: Other: MRI examinations
- head and neck cancer or thyroid cancers (differentiated and undifferentiated): All patients, irrespective of treatment regimen, will be imaged on a 1.5T or 3T MR scanner prior to treatment initiation. Follow up imaging for patients undergoing surgery only will be as per clinical standard of care and not on this protocol. Patients undergoing treatment in radiation oncology and/or medicine will have imaging studies during week 2 of treatment. If patients receive 70Gy, they will also receive a scan during week 4 of treatment, if needed by treating physician. Scans will be performed to derive MRI biomarkers indicative of therapeutic mechanisms of action or efficacy will also be performed.
  Interventions: Other: MRI examinations

INTERVENTIONS:
Other: MRI examinations — Patients will be imaged on a 1.5 T or 3 T MR scanner either from GE or Philips. Patients will receive a test-retest scan in on session prior to start of treatment. Patients who will be receiving radiation therapy treatment at main campus, will also be imaged weekly during their course of treatment.
  Groups: recurrent or metastatic head and neck cancer patients
Other: MRI examinations — Patients will be imaged on a 1.5 T or 3T MR scanner within one week prior to treatment initiation and at two months and four months after treatment completion (+/- 1 week).
  Groups: head and neck cancer or thyroid cancers (differentiated and undifferentiated)

SUMMARY:
Magnetic resonance imaging (MRI) is a diagnostic technique that takes pictures of organs of the body. It uses magnetic fields and radio waves that cannot be felt. This makes specific organs, blood vessels, or tumors easier to see. Diffusion MRI lets us measure the motion of water in the tumor.

The purpose of this study is to see if new MRI methods can give us more information about the tumor.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Group 1 patients: Presence of a suspicious metastatic lesion or suspicious for recurrent disease in the head and neck region.
* Group 2 patients:

  * Biopsy proven recurrent or metastatic or definitive head and neck cancer or (differentiated and undifferentiated) thyroid cancers in the head and neck region only.
  * Patients planning to undergo reatment at MSK

Exclusion Criteria:

* Patient would require anesthesia for the study
* Patients who are claustrophobic
* Patients selecting treatment outside of MSK
* Known reaction to Gd based contrast agent
* Patients who have presence of a known contradiction to MRI

  * Pacemaker
  * Aneurysm clips
  * Patients with implants that are contradicted for MR imaging will be excluded
  * Pregnant
  * Age and mental status wherein he /she is unable to cooperate for MRI study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MSK clinics in the medicine, surgery and radiation oncology departments.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-03-16 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
For group 1: number of patients that have biomarkers that maybe early response to therapy indicators | 1 year
  The study is designed to determine if the MRI will provide quantitative imaging biomarkers to predict or assess early treatment response in R/M head and neck cancers. The MR data will be compared with clinical follow-up data. Additional sequence parameters.
For group 2: number of patients response to treatment | 1 year
  will be assessed using ROC curves with RECIST with the RECIST version 1.1 response as the gold standard and change in DW-MRI and image feature metrics as predictors.

CONTACTS AND LOCATIONS:
Overall Officials: Amita Dave, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm